CLINICAL TRIAL: NCT04785417
Title: Effect of Touch Screen Tablet on Fine Motor Function un Children With Hemiparetic Cerebral
Brief Title: Effect of Touch Screen Tablet on Fine Motor Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, hanaa mohsen, lecturer in the department of paediatrics and paediatric surgery , faculty of physical therapy, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HANA 6
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Hemiplegic Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): received conventional occupational therapy program
- STUDY GROUP (Experimental): received conventional occupational therapy program in addition to using tablet
  Interventions: Other: touch screen tablet

INTERVENTIONS:
Other: touch screen tablet — traditional occupational therapy in addition to games on tablet
  Arms: STUDY GROUP

SUMMARY:
the objective of this study to asses the effect of touch screen tablet on fine motor functions

ELIGIBILITY:
Inclusion Criteria:

* hemiplegia
* mid spasticity of upper limb
* able to follow instructions

Exclusion Criteria:

* fixed deformities visual or respiratory problem

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
pinch gauge | pre and post three month of intervention increase score indicate improvement
  used to asses pinch strength
QUEST | pre and post three month of intervention increase score indicate improvement
  to asses the fine motor function
nine hole pegboard test | pre and post three month of intervention increase score indicate improvement
  used to asses the fine motor function

CONTACTS AND LOCATIONS:
Overall Officials: hanaa mohsen, Principal Investigator — lecturer ,faculty of physical therapy, Badr universality in Cairo
Locations (1):
- Hanaa Mohsen, Cairo, Egypt